CLINICAL TRIAL: NCT07143526
Title: Comparison of Two Swept-source Optical Coherence Tomography Angiography (OCTA) Devices (Bmizar and Plexelite) for Detecting Macular Neovascularisation With Large (More Than 250 Microns) Pigment Epithelium Detachment (PED) in Age Related Macular Degeneration
Brief Title: Comparison of the Sensibility of Swept Source Optical Coherence Tomography Devices in the Detection of Neovascularisation in Large Pigment Epithelium Detachments
Status: Not yet recruiting | Type: Observational
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Marco Rocco Pastore, Department of Ophtalmology Clinical Assistant, University of Trieste
Other Study IDs: 1030725
Record Dates: First submitted 2025-08-11; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: AMD - Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography Angiography (OCT-A) — Two Optical Coherence Tomography Angiography swept source devices are compared for the detection of large pigment epithelium detachments in age related macular degeneration. The sensitivity of the devices is compared in both the automatic segmentation done by the device and the manual segmentation done by a retina specialist.

SUMMARY:
The goal of this observational study is to compare swept source optical coherence tomography devices ability to detect macular neovascularisation when there is a large pigment epithelium detachment higher than 250 microns

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for neovascular age related macular degeneration (AMD)
* Presence of a pigmentary epithelium detachment higher than 250 microns measured on structural optical coherence tomography (OCT)

Exclusion Criteria:

* Poor image quality or signal strength
* Undefined retina layers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated for neovascular age related macular degeneration (AMD)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the detection of neovascularisation in large pigment epithelium detachment by swept source optical coherence tomography devices | Day 1
  The optical coherence tomography angiography devices are known to have a difficult time detecting neovascularisation in the cases of large pigment epithelium detachments (PED), because of the many layers and the distance the OCT signal has to cross. The automatic retina segmentation (done by the device of the different retina layers plays a big role in this detection. It's also disturbed by the height of the PED.
  This study aims to compare the sensitivity of two swept source OCT devices available in the market : Bmizar, Towardpi and Plexelite, Zeiss.
  After the exam image acquisition, a retina specialist will try to make a manual segmentation of the retina analysed to help the detection of macular neovascularisation that would have been missed in the "normal" automatic segmentation done by the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No